CLINICAL TRIAL: NCT01625182
Title: A Double-blind, Randomized, Multicenter, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Fingolimod 0.5 mg Administered Orally Once Daily Versus Placebo in Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Brief Title: Evaluate Efficacy and Safety of Fingolimod 0.5 mg Orally Once Daily Versus Placebo in Chronic Inflammatory Demyelinating Polyradiculoneuropathy Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CFTY720I2201; 2011-005280-24 (EudraCT Number)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-09

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Keywords: chronic inflammatory demyelinating polyradiculoneuropathy, CIDP, FTY720, fingolimod.
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fingolimod (FTY720) (Experimental): Participants received Fingolimod 0.5 mg orally once daily.
  Interventions: Drug: Fingolimod
- Placebo (Placebo Comparator): Participants received matching placebo to Fingolimod orally once daily.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Fingolimod — Fingolimod 0.5 mg capsules
  Arms: Fingolimod (FTY720)
Drug: Placebo Comparator — Matching placebo capsules
  Arms: Placebo

SUMMARY:
The study was designed to evaluate the efficacy and safety of fingolimod in the treatment of chronic inflammatory demyelinating polyradiculoneuropathy compared with placebo.

DETAILED DESCRIPTION:
This study was a double-blind, randomized, multicenter, placebo-controlled, parallel-group study in patients with a diagnosis of chronic inflammatory demyelinating polyradiculoneuropathy and treated with IVIg, corticosteroids, or both therapies prior to study entry. Patients meeting the eligibility criteria were randomly assigned in a ratio of 1:1 to receive oral fingolimod (0.5 mg/day) or matching placebo.

The study consisted of 3 periods: a Screening Period, a Double-blind Treatment Period and a Follow-up Period after discontinuation of study drug treatment. Patients who complete the study will have an option to enter an extension.

ELIGIBILITY:
Inclusion Criteria

* written informed consent must be obtained before any assessment is performed
* The diagnosis of CIDP will use the definition of the EFNS/PNS Task Force First Revision. Patients must either have a clinical diagnosis of CIDP fulfilling the clinical inclusion criteria for typical CIDP or one of the following atypical forms of CIDP: pure motor, or asymmetrical (MADSAM [Lewis-Sumner syndrome]), or IgA or IgG (not IgM) MGUS paraprotein associated.
* All patients must also fulfill the clinical exclusion criteria and the definite electrodiagnostic criteria of the EFNS/PNS Task Force First Revision.
* disability defined by an INCAT Disability Scale score of 1-9 or, if INCAT score is 0, a documented history of disability sufficient to require treatment within the past 2 years following reduction or interruption of CIDP treatment
* receiving IVIg treatment (minimal dose equivalent to 0.4 g/kg every 4 weeks for a minimum of 12 weeks) or corticosteroids (minimal dose equivalent to prednisone 10 mg/day) treatment prior to the screening visit
* history of documented clinically meaningful deterioration confirmed by clinical examination during therapy or upon interruption or reduction of therapy within 18 months prior to Screening
* stable CIDP symptoms for the 6 weeks before randomization

Exclusion Criteria

* other chronic demyelinating neuropathies, including: Distal Acquired Demyelinating Symmetric Neuropathy (DADS) Multifocal Motor Neuropathy (MMN) pure sensory CIDP hematopoietic malignancy except for MGUS
* conditions in which the pathogenesis of the neuropathy may be different from CIDP such as: Lyme disease, POEMS syndrome, osteosclerotic myeloma, Castleman's disease
* treatment with plasma exchange within 2 months of randomization, immunosuppressive/chemotherapeutic medications: azathioprine, cyclophosphamide, cyclosporine, mycophenolate, etanercept, methotrexate tacrolimus or other immunosuppressive drugs within 6 months of randomization or 5 half-lives (whichever is later), Rituximab in the 2 years prior to randomization (patients that have received rituximab between 1 and 2 years should have B-cell levels within normal range), other cytotoxic immunosuppressive medications with sustained effects (including mitoxantrone, alemtuzumab, cladribine) at any time, hematopoietic stem cell transplantation at any time

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-12-22 (Actual); Primary Completion 2016-09-03 (Actual); Study Completion 2016-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (66):
- United States (12):
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Patchogue, New York
  - Novartis Investigative Site, Plainview, New York
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Burlington, Vermont
- Australia (4):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Canada (4):
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Greenfield Park
  - Novartis Investigative Site, Montreal
- Novartis Investigative Site, Prague, Czechia
- France (6):
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Strasbourg
- Germany (5):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Göttingen
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (7):
  - Novartis Investigative Site, Legnano, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Cefalù, PA
  - Novartis Investigative Site, Ferrara
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Rome
- Japan (6):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Aomori, Aomori
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Bunkyo, Tokyo
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Chiba
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Maastricht
- Poland (3):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Lodz
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid
- United Kingdom (5):
  - Novartis Investigative Site, Headington, Oxfordshire
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hughes R, Dalakas MC, Merkies I, Latov N, Leger JM, Nobile-Orazio E, Sobue G, Genge A, Cornblath D, Merschhemke M, Ervin CM, Agoropoulou C, Hartung HP; FORCIDP Trial Investigators. Oral fingolimod for chronic inflammatory demyelinating polyradiculoneuropathy (FORCIDP Trial): a double-blind, multicentre, randomised controlled trial. Lancet Neurol. 2018 Aug;17(8):689-698. doi: 10.1016/S1474-4422(18)30202-3. Epub 2018 Jul 9. PMID 30001923

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned randomly to each treatment group in a 1:1 ratio.
Period: Overall Study
Arm/Group | Fingolimod (FTY720) | Placebo
Started | 54 | 52
Completed | 34 | 41
Not Completed | 20 | 11
Not completed — Administrative problems | 1 | 0
Not completed — Protocol deviation | 0 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lack of Efficacy | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod (FTY720) | Placebo | Total
Number analyzed (Participants) | 54 | 52 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (13.32) | 54.6 (11.68) | 54.5 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 37 | 30 | 67

OUTCOME MEASURES:

1. Primary Outcome: Time to First Confirmed Worsening on the Adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Scale
Description: Confirmed worsening in CIDP was measured by the adjusted INCAT Disability Scale. The adjusted INCAT disability scale measures arm disability and leg disability. For arm disability the scale ranges from 0 (no upper limb problems) to 5 (inability to use either arm for any purposeful movement). The leg disability scale ranges from 0 (walking not affected) to 5 (restricted to wheelchair, unable to stand and walk a few steps with help). The total adjusted INCAT disability score is calculated by the sum of the arm and leg disability scores where the total score ranges from 0 to 10. A confirmed worsening was defined as an increase by 1 or more points on the adjusted INCAT disability scale from the value at baseline.
Time Frame: Month 12
Population: The full analysis set, which included all participants who were assigned randomly to receive treatment, was analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fingolimod (FTY720) | Placebo
Number analyzed (Participants) | 54 | 52
Days | 721.0 [159.0 to NA] — The 95% upper confidence interval not estimable. | 540.0 [183.0 to NA] — The 95% upper confidence interval not estimable.
Statistical Analysis 1: Comparison: Fingolimod (FTY720) vs Placebo; Test type: Superiority or Other; p = 0.9838, Regression, Cox; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.6 to 1.7]

2. Secondary Outcome: Change From Baseline for Grip Strength, Dominant Hand
Description: Grip strength measurements were done using a vigorimeter. With this device, the pressure in the bulb exercised by the participant was registered on a manometer via a rubber junction tube. Both the dominant and non-dominant hands were tested. A negative change from baseline indicates deterioration.
Time Frame: baseline, Month 6, Month 12
Population: Only participants from the FAS, who had non-missing baseline values and the given post-baseline values, were included in the analysis. The FAS included all participants who were assigned randomly to receive treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Fingolimod (FTY720) | Placebo
Number analyzed (Participants) | 53 | 50
kPa
  Month 6 | -2.6 [-8.09 to 2.80] | -3.8 [-9.37 to 1.70]
  Month 12 | -0.8 [-6.47 to 4.96] | -3.9 [-9.68 to 1.94]

3. Secondary Outcome: Change From Baseline for Grip Strength, Non-dominant Hand
Description: as for outcome 2
Time Frame: baseline, Month 6, Month 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Fingolimod (FTY720) | Placebo
Number analyzed (Participants) | 53 | 50
kPa
  Month 6 | -2.7 [-8.13 to 2.66] | -6.1 [-11.59 to -0.66]
  Month 12 | -1.2 [-6.69 to 4.37] | -5.0 [-10.57 to 0.64]

4. Secondary Outcome: Change From Baseline for Rasch-Built Linearly Weighted Overall Disability Scale (R-ODS)
Description: This questionnaire was constructed using the patients' perception of their ability to perform daily and social activities. The questionnaire comprises 24 items ranging from ability to read a book or newspaper (as the easiest item to accomplish) to ability to run (most difficult item to accomplish). The obtained raw summed score was translated subsequently to a convenient centile metric score ranging from 0 (most severe disability) to 100 (no disability at all). A higher score indicated a better health status. A negative change from baseline indicates deterioration.
Time Frame: baseline, Month 6, Month 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fingolimod (FTY720) | Placebo
Number analyzed (Participants) | 54 | 51
score on a scale
  Month 6 | -6.4 [-9.57 to -3.15] | -5.5 [-8.89 to -2.21]
  Month 12 | -5.7 [-9.07 to -2.37] | -5.1 [-8.54 to -1.57]

ADVERSE EVENTS:
Arm/Group | Fingolimod (FTY720) | Placebo | Overall Participants
Serious Adverse Events (participants affected / at risk) | 9/54 | 4/52 | 13/106
Other Adverse Events (participants affected / at risk) | 40/54 | 42/52 | 82/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (FTY720) (N=54) | Placebo (N=52) | Overall Participants (N=106)
Oedema peripheral (General disorders) | 1 | 0 | 1
Abdominal sepsis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 1 | 1
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 2 | 1 | 3
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (FTY720) (N=54) | Placebo (N=52) | Overall Participants (N=106)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 2 | 2
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 3 | 6
Cushingoid (Endocrine disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Blepharitis (Eye disorders) | 2 | 0 | 2
Cataract (Eye disorders) | 1 | 3 | 4
Diplopia (Eye disorders) | 0 | 1 | 1
Eye pain (Eye disorders) | 1 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 1
Iritis (Eye disorders) | 0 | 1 | 1
Macular oedema (Eye disorders) | 1 | 1 | 2
Meibomianitis (Eye disorders) | 1 | 0 | 1
Metamorphopsia (Eye disorders) | 0 | 1 | 1
Retinal disorder (Eye disorders) | 0 | 1 | 1
Retinoschisis (Eye disorders) | 1 | 0 | 1
Subretinal fluid (Eye disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 2 | 0 | 2
Visual acuity reduced (Eye disorders) | 1 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 1
Vitreous detachment (Eye disorders) | 1 | 1 | 2
Vitreous floaters (Eye disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 3
Change of bowel habit (Gastrointestinal disorders) | 1 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Gingival cyst (Gastrointestinal disorders) | 0 | 1 | 1
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 6 | 8
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 1
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 1
Discomfort (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 4 | 6 | 10
Influenza like illness (General disorders) | 1 | 1 | 2
Local swelling (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Pain (General disorders) | 1 | 1 | 2
Peripheral swelling (General disorders) | 1 | 1 | 2
Pyrexia (General disorders) | 2 | 1 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 2
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 3 | 1 | 4
Candida infection (Infections and infestations) | 1 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 2 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Ear infection (Infections and infestations) | 1 | 0 | 1
Folliculitis (Infections and infestations) | 2 | 3 | 5
Gastroenteritis (Infections and infestations) | 0 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 2
Herpes zoster (Infections and infestations) | 1 | 1 | 2
Influenza (Infections and infestations) | 2 | 0 | 2
Laryngitis (Infections and infestations) | 1 | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 6 | 7 | 13
Onychomycosis (Infections and infestations) | 0 | 1 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 1
Parasitic gastroenteritis (Infections and infestations) | 0 | 1 | 1
Periodontitis (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 2
Tinea cruris (Infections and infestations) | 0 | 1 | 1
Tinea infection (Infections and infestations) | 1 | 0 | 1
Tonsillitis bacterial (Infections and infestations) | 1 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3
Urinary tract infection (Infections and infestations) | 3 | 1 | 4
Vulvovaginal candidiasis (Infections and infestations) | 1 | 1 | 2
Wound infection (Infections and infestations) | 1 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 1 | 5
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1 | 3
Amylase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 1
Blood urine present (Investigations) | 1 | 0 | 1
Carbon monoxide diffusing capacity decreased (Investigations) | 1 | 0 | 1
Cardiac murmur (Investigations) | 1 | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 3
Glycosylated haemoglobin increased (Investigations) | 1 | 1 | 2
Grip strength decreased (Investigations) | 1 | 0 | 1
Heart rate increased (Investigations) | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0 | 2
Hepatitis A virus test positive (Investigations) | 1 | 0 | 1
Occult blood (Investigations) | 0 | 1 | 1
Optic nerve cup/disc ratio increased (Investigations) | 0 | 1 | 1
Pulmonary function test decreased (Investigations) | 0 | 1 | 1
Serum ferritin decreased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 3 | 10
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1 | 1
Coordination abnormal (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 2 | 5
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 12 | 8 | 20
Hypoaesthesia (Nervous system disorders) | 2 | 2 | 4
Memory impairment (Nervous system disorders) | 1 | 1 | 2
Meningism (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 5 | 0 | 5
Parkinsonism (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 2 | 1 | 3
Somnolence (Nervous system disorders) | 1 | 2 | 3
Syncope (Nervous system disorders) | 2 | 1 | 3
Tremor (Nervous system disorders) | 1 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 4 | 5
Irritability (Psychiatric disorders) | 0 | 1 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0 | 1
Breast cyst (Reproductive system and breast disorders) | 1 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 1
Breast swelling (Reproductive system and breast disorders) | 0 | 1 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Chloasma (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Lentigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Hot flush (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 10 | 1 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.